CLINICAL TRIAL: NCT07103538
Title: The Effect of the Reflective Practices on Nursing Students' Empathy and Compassion Levels: A Randomized Controlled Trial
Brief Title: The Effect of the Reflective Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Fatma DURSUN ERGEZEN, Assistant Professor, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FErgezen
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Empathy; Compassion; Nursing Student
Keywords: empathy; compassion; reflective practices

STUDY DESIGN:
Masking Description: The statistician was masked in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention was implemented as part of a nursing course consisting of 4 hours of theoretical instruction, 4 hours of laboratory practice, and 8 hours of clinical practice. For 14 weeks, reflective practice was integrated into both the laboratory and clinical components. In the laboratory sessions, clinical scenarios were developed based on five common topics (e.g., infection control, vital signs) that students are likely to encounter during clinical practice. Students performed these scenarios by taking on different roles. Following each role-play, structured reflection sessions were conducted with the students. In the clinical setting, the final hour of each practice day was allocated for reflection. After completing an online reflection form, students had the opportunity to engage in group discussions if they wished to reflect further.
  Interventions: Behavioral: Reflective practices
- Control (No Intervention): Students followed the same laboratory and clinical curriculum but did not participate in any structured reflective practices. They received standard instruction in psychomotor skills and routine clinical procedures without the inclusion of role-play, scenario-based learning, or debriefing sessions.

INTERVENTIONS:
Behavioral: Reflective practices — The intervention was implemented as part of a nursing course consisting of 4 hours of theoretical instruction, 4 hours of laboratory practice, and 8 hours of clinical practice. For 14 weeks, reflective practice was integrated into both the laboratory and clinical components. In the laboratory sessions, clinical scenarios were developed based on five common topics (e.g., infection control, vital signs) that students are likely to encounter during clinical practice. Students performed these scenarios by taking on different roles. Following each role-play, structured reflection sessions were conducted with the students. In the clinical setting, the final hour of each practice day was allocated for reflection. After completing an online reflection form, students had the opportunity to engage in group discussions if they wished to reflect further.
  Arms: Intervention

SUMMARY:
The aim of this study was to explore the effects of reflective practices on nursing students' empathy and compassion levels.

Hypothesis H1-1: Reflective practices affect nursing students' empathy level. H1-2: Reflective practices affect nursing students' compassion level.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Enrollment in the "Fundamentals of Nursing-II" course
* Taking the course for the first time
* Not having previously received training in reflective practice
* Being registered in Class B

Exclusion Criteria:

* Refusal to participate in the study at any stage of the study process
* Failure to fully complete the data collection forms

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Empathy | Data were collected at two different time points: At recruitment (T0) and in the 14th week (T1)
  The Jefferson Scale of Empathy for Nursing Students was designed to measure empathy levels in nursing students. The Turkish adaptation consists of 18 items across the same three sub-dimensions. The scale is based on a 7-point Likert-type format (1 = Strongly disagree to 7 = Strongly agree), yielding a total score ranging from 18 to 126. Higher total scores reflect greater levels of empathy.
Compassion | Data were collected at two different time points: At recruitment (T0) and in the 14th week (T1)
  The Compassion Scale comprises 24 items and six subscales: kindness, indifference, common humanity, separation, mindfulness, and disengagement. The subscales of indifference, disengagement, and separation are reverse-scored prior to calculating the overall compassion score. Total scores range from 24 to 120, with higher scores indicating higher levels of compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Durkin M, Gurbutt R, Carson J. Effectiveness of an online short compassion strengths course on nursing students compassion: A mixed methods non-randomised pilot study. Nurse Educ Today. 2022 Apr;111:105315. doi: 10.1016/j.nedt.2022.105315. Epub 2022 Feb 26. PMID 35290862
- [Background] Dreifuerst KT. Using debriefing for meaningful learning to foster development of clinical reasoning in simulation. J Nurs Educ. 2012 Jun;51(6):326-33. doi: 10.3928/01484834-20120409-02. Epub 2012 Apr 9. PMID 22495923
- [Background] Contreras JA, Edwards-Maddox S, Hall A, Lee MA. Effects of Reflective Practice on Baccalaureate Nursing Students' Stress, Anxiety and Competency: An Integrative Review. Worldviews Evid Based Nurs. 2020 Jun;17(3):239-245. doi: 10.1111/wvn.12438. Epub 2020 Apr 24. PMID 32329238
- [Background] Coleman D, Willis DS. Reflective writing: the student nurse's perspective on reflective writing and poetry writing. Nurse Educ Today. 2015 Jul;35(7):906-11. doi: 10.1016/j.nedt.2015.02.018. Epub 2015 Mar 14. PMID 25802097
- [Background] Arman M. Empathy, sympathy, and altruism-An evident triad based on compassion. A theoretical model for caring. Scand J Caring Sci. 2023 Sep;37(3):862-871. doi: 10.1111/scs.13163. Epub 2023 Mar 21. PMID 36942653
- [Background] Adamson E, Dewar B. Compassionate Care: Student nurses' learning through reflection and the use of story. Nurse Educ Pract. 2015 May;15(3):155-61. doi: 10.1016/j.nepr.2014.08.002. Epub 2014 Sep 19. PMID 25754833